CLINICAL TRIAL: NCT03273101
Title: Does Self-initiated Sit-to-stand Training With Assistive Device Regain the Independence of Sit-to-stand in Stroke Patient? A Single-blinded Randomised Controlled Trial.
Brief Title: Sit-to-stand Training in Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tai Po Hospital (Other Government)
Responsible Party: Principal Investigator, Ng Chee Man, Joey, Principal investigator, Tai Po Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014.427
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The sit-to-stand training is assisted by mechanical device
  Interventions: Device: Mechanical assisted sit-to-stand training group
- Control group (Active Comparator): The sit-to-stand training is assisted by manual device
  Interventions: Other: Manual assisted sit-to-stand training group

INTERVENTIONS:
Device: Mechanical assisted sit-to-stand training group — Mechanical assisted sit-to-stand training 100 repetitions or 10 mins / session 10 sessions
  Other Names: sit-to-stand trainer
  Arms: Intervention group
Other: Manual assisted sit-to-stand training group — Manual assisted sit-to-stand training 100 repetitions or 10 mins / session 10 sessions
  Other Names: physiotherapist assisted
  Arms: Control group

SUMMARY:
Background: It is unknown whether the self-initiated sit-to-stand training with assistive device is effective to regain the independence of sit-to-stand in stroke patients.

Objective: To compare the effectiveness of self-initiated sit-to-stand training by assistive device, with manual sit-to-stand training.

Design: Parallel randomised controlled and assessor blinded trial between Jan 2015 and May 2018. Randomisation was performed by drawing lots to allocate treatment to patient.

Setting: A rehabilitation hospital in Hong Kong

Participants: 69 patients in medical wards with unilateral hemiparetic stroke. 52 patients fulfilled the study requirements.

Intervention: Ten sessions of intervention with conventional physiotherapy program followed, by self-initiated sit-to-stand training with assistive device, or by manual sit-to-stand training.

Main outcome measure: Number of patients regained the independence of sit-to-stand, Sit-to-stand test from the balance master® and Five-repetitions sit-to-stand test.

Results: 69 patients (intervention n=36; control n=33) were randomized (mean age 69.8 (SD, 10.6), mean post stroke days 18.6 (SD 16.0)) for intention to treat analysis. 17 patients were excluded because of dropout before 10 sessions of training, leaving 52 (n=26; n=26) patients for per protocol analysis. 18 patients in intervention group and 10 patients in control group had regained the independence of sit-to-stand (Phil and Cramer's V: -0.31 and 0.31). The patients in intervention group were faster to complete the Five-repetition sit-to-stand test than the control group (32.7 secs (SD, 1.93) v 48.4 secs (SD, 6.8); 95% confidence interval, -30.8 to -0.7; p<0.05). No adverse side effects occurred during and after the training across groups.

Conclusions: Self-initiated sit-to-stand training by assistive device can help more stroke patients regain the independence of sit-to-stand.

ELIGIBILITY:
Inclusion Criteria:

* first episode of unilateral stroke with hemiparesis,
* able to understand and follow simple verbal instructions,
* able to sit unsupported for at least two minutes
* require lifting assistance to stand up from a 18 inches high plinth

Exclusion Criteria:

* severe pain in the lower extremities when weight bearing or performing movement
* any other acute comorbid diseases such as unstable angina, recent myocardial infarction
* unstable medical / psychological condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Number of patients regained the independence of sit-to-stand | After 10 sessions of training
  To compare how many patients can regain the independence of sit-to-stand between groups
Sit-to-Stand Test (SST) from the Balance Master® | After 10 sessions of training
  To assess the quality of sit-to-stand of patient
Five-Repetition Sit-to-Stand Test | After 10 sessions of training
  To assess the functional strength of lower limb, balance and transition move of patient

CONTACTS AND LOCATIONS:
Overall Officials: Ng Chee Man, Joey, Master, Principal Investigator — Tai Po Hospital; Woo Ka Ho, Marc, Master, Study Director — Prince of Wales Hospital

IPD SHARING:
Plan to Share IPD: No